CLINICAL TRIAL: NCT03455153
Title: The Association of Physical Activity Levels and Inflammatory Markers in COPD Patients Following Pulmonary Rehabilitation
Brief Title: Association of Physical Activity Levels and Inflammatory Markers Following Pulmonary Rehabilitation
Acronym: PALI-COPD
Status: Completed | Type: Observational
Sponsor: University of Lincoln (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 18/WM/0081
Record Dates: First submitted 2018-02-07; First posted 2018-03-06 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: COPD
Keywords: Pulmonary Rehabilitation; Neutrophils
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples will be used on the day of collection and analysed before being appropriately disposed of on the same day. Blood samples will be centrifuged with separated acellular plasma to be frozen at -80c for later analysis of cellular content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Most active: COPD patients with higher physical activity levels as defined by daily step counts.
  Interventions: Other: Physical activity monitoring
- Least active: COPD patients with lower physical activity levels as defined by daily step counts.
  Interventions: Other: Physical activity monitoring

INTERVENTIONS:
Other: Physical activity monitoring — COPD patients will wear an accelerometer and complete questionnaires related to daily physical activity levels for 7 days before returning for a clinic visit.

SUMMARY:
COPD is characterised by irreversible airflow limitation that is usually progressive and associated with an enhanced chronic inflammatory response. This inflammation can be amplified with flare-ups that are commonly seen in COPD patients. Pulmonary rehabilitation is one of the most effective methods of managing chronic obstructive pulmonary disease (COPD). Pulmonary rehabilitation has been seen to induce improvements in functional capacity and quality.

In healthy individuals, exercise has been shown to induce an anti-inflammatory response when performed regularly. However, the effects of exercise on inflammation in COPD are unclear. Our initial CIMPRES-COPD study has looked into the effects of short-term exercise, as part of pulmonary rehabilitation, on inflammation. However, this trial will examine the inflammatory response in COPD patients who are most active following pulmonary rehabilitation against those who are least active.

This study will split participants into 2 groups according to physical activity level following pulmonary rehabilitation. We will recruit 40 COPD patients who provided a sample in the initial CIMPRES-COPD study to explore inflammatory responses in those who are most active and least active. By better understanding the mechanisms of how long-term physical activity levels affects inflammation in COPD, we could design better interventions to increase physical activity levels following pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with any severity of COPD (according to British Thoracic Society criteria, i.e. >10 pack year smoking history and post bronchodilator spirometry FEV1/FVC ratio <0.70 and FEV<80%)
* Previously enrolled on pulmonary rehabilitation providing at least one sample for the CIMPRES-COPD trial.

Exclusion Criteria:

* Any unstable ongoing cardiovascular events.
* Other active inflammatory conditions (e.g. rheumatoid arthritis, cancer).
* Known asthma, allergic rhinitis or other respiratory disease (bronchiectasis, pulmonary fibrosis).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients who have enrolled on pulmonary rehabilitation and took part in the initial CIMPRES-COPD study.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Cytokines | May 2018 - August 2018
  Changes in concentration of inflammatory cytokines in the plasma of all participants using ELISA's (mg/L)

SECONDARY OUTCOMES:
Leukocyte count | May 2018 - August 2018
  Changes in total and differential leukocyte count in all participants (10^9.L-1)
Cell function | May 2018 - August 2018
  Changes in function of the following cells: myeloperoxidase, neutrophil elastase, MMP-8, MMP-9, TNF-a in the plasma of all participants using ELISA's (mg/L)
Cell sensitivity to corticosteroids | May 2018 - August 2018
  Changes in cell sensitivity to corticosteroids and forskolin in all participants (expressed as fold increase from not treated samples)

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Lindum Medical Practice, Lincoln, Lincolnshire
  - Nettleham Medical Practice, Lincoln, Lincolnshire
  - Birchwood Medical Practice, Lincoln, Lincolnshire

IPD SHARING:
Plan to Share IPD: No